CLINICAL TRIAL: NCT01607216
Title: Prematurity and Respiratory Outcome Program: Single Center Study of Functional and Lymphocytic Markers of Respiratory Morbidity in Hyperoxic Preemies
Brief Title: Functional and Lymphocytic Markers of Respiratory Morbidity in Hyperoxic Preemies
Status: Completed | Type: Observational
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH); University at Buffalo (Other)
Responsible Party: Principal Investigator, Gloria Pryhuber, Professor, University of Rochester
Other Study IDs: 37933; U01HL101813 (NIH)
Record Dates: First submitted 2012-03-14; First posted 2012-05-30 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Prematurity; Symptomatic Respiratory Disease; Bronchopulmonary Dysplasia
Keywords: Prematurity; Respiratory Illness; Lung Function; Lung Disease
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Several types of biospecimens are to be collected:
  Cord Blood Tracheal Aspirates Urine Stool Saliva Blood
  DNA collection is optional.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Premature Infant: Infants born 23 0/7 weeks gestation to 35 6/7 weeks gestation.
- Healthy Full Term Infants: Infants born between 37 0/7 weeks gestation to 41 6/7 weeks gestation.

SUMMARY:
This is an observational study that proposes to collect clinical, physiological, cellular and molecular information in an attempt to identify a set of factors that may predict the risk for persistent lung disease in babies born prematurely.

DETAILED DESCRIPTION:
Approximately 550,000 babies born prematurely each year in the United States suffer from birth at a time in development when the respiratory tract and immune system would normally be protected and maintained in a naïve state. This project is a component of the NIH Prematurity and Respiratory Outcomes Program (PROP) whose goals are the identification of disease mechanisms and biomarkers to stratify premature infants, at the time of discharge, for their risk of subsequent pulmonary morbidity. This Clinical Research Center (CRC) project will investigate prematurity-dependent alterations in cellular innate and adaptive immune systems resulting in increased susceptibility to respiratory infections and environmental irritants, and leading to respiratory morbidity in the first year of life. Prior studies have established developmental (maturity) and disease-related changes in circulating and pulmonary lymphocyte populations but a comprehensive assessment of their relationship to disease risk/outcome has not been undertaken. We hypothesize that cellular and molecular immuno-maturity is altered due to intrinsic and extrinsic factors presented by premature birth in such a way as to reduce resistance to viral infections and to promote cytotoxic damage to the lung. We will evaluate immunologic maturity by comprehensively phenotyping lymphocyte populations in peripheral blood sampled at premature delivery, at the time of discharge from the hospital and at twelve months corrected age. The lymphocytic phenotype will be analyzed particularly in the context of gestational age and maternal-fetal stressors capable of modulating oxidative stress (oxygen exposure, infection and environmental tobacco smoke exposure). Additionally, we will assess changes in the molecular phenotype of isolated CD8 lymphocytes, a cell type preferentially recruited to the lungs of premature infants and capable of contributing to disease pathogenesis, by genome-wide expression profiling, in order to uncover novel disease pathways and define a gene expression signature associated with disease risk. Finally, we propose to build a statistical model, using cellular and molecular phenotypes and additional clinical variables, for stratifying risk of lung morbidity within the first year of life.

ELIGIBILITY:
Inclusion Criteria:

1. Premature infants born at gestational age 24 0/7 to 35 6/7 week and admitted to the Neonatal Intensive Care Unit or normal newborn nursery at URMC or UB
2. Healthy term infants 37 0/7 to 41 6/7 recruited from the birthing centers or Ob/Gyn floors (3-1200 at URMC) prior to discharge
3. Infants who are less than or equal to 7 days old

Exclusion Criteria:

1. The infant is not considered to be viable (therapies limited due to futility decision made by clinical care team)
2. Congenital heart disease (not including PDA and hemodynamically insignificant VSD or ASD)
3. Structural abnormalities of the upper airway, lungs or chest wall
4. Other congenital malformations or syndromes that adversely affect life expectancy or cardio-pulmonary development
5. Family is unlikely to be available for long-term follow-up as determined by the site investigators dependent on the distance of the infant's residence from the follow-up center and/or family plans to move out of the region
6. Family does not speak or understand English

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Eligible subjects are limited to patients born at the Golisano Children's Hospital at the University of Rochester Medical Center and at Women's and Children's Hospital, University at Buffalo. All admissions to the participating Neonatal Intensive Care Units will be screened for eligibility.
Sampling Method: Non-Probability Sample
Enrollment: 277 (Actual)
Dates: Start 2011-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Symptomatic Respiratory Disease (SRD) | Assessed every three months until 1 year corrected gestational age
  The primary goal of the PROP studies (single center and multicenter protocols) is to identify biomarkers (biochemical, physiological and genetic) and clinical variables that are associated with and thus potentially predictive of pulmonary status in preterm infants up to 1 year corrected age. We propose a composite primary outcome of SRD that is based on serial parental reports of respiratory symptoms, medications, hospitalizations and dependence on technology during the first year of life.

SECONDARY OUTCOMES:
Assessment of T lymphocyte numbers, subsets (CD4, CD8) and functional phenotype determined by flow cytometry. | Measured and compared at birth, at term corrected gestational age and at 1 year corrected gestational age
  Assessment of T lymphocyte numbers, subsets (CD4, CD8) and functional phenotype including characteristics of effector and memory function, and intracellular cytokine production in response to in vitro T cell receptor nonspecific and specific stimulation
Measure of severity of lung disease at 40 +/- 5 weeks corrected gestational age | From birth at premature gestational age to at 40 +/- 5 weeks corrected gestational age
  Severity of lung disease will be assessed by length of time on mechanical ventilation, length of time on oxygen, oxygen requirement at 36 weeks corrected gestational age, need for pulmonary medications at determined at hospital discharge, or at 40 +/- 5 weeks corrected gestational age.
Statistical correlation of CD4 and CD8 lymphocyte function with severity and persistence of lung disease. | At at 40 +/- 5 weeks corrected gestational age and at one year of age
  The severity of lung disease prior to first hospital discharge and the persistence and severity of SRD in the first year of life will be compared with the T cell lymphocyte phenotypes at birth, at hospital discharge and at one year of life. Specifically, at minimum, the ability of T lymphocytes at rest and after stimulation to produce interferon gamma at the test time points will be compared with the history of lung disease. The intent is to identify biomarkers and to suggest immune-mediated mechanisms for lung disease in preterm infants
Gene expression analysis of CD8 cells collected by FACS from preterm infants nearing discharge | At 40 +/- 5 weeks corrected gestational age
  Patterns of gene expression identified in isolated and sorted CD8 T cells from preterm infants just prior to discharge from the neonatal intensive care unit will be identified and compared to the severity and persistence of symptomatic respiratory disease (SRD) over the first year of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Pryhuber, MD, Principal Investigator — University of Rochester; Rita Ryan, MD, Principal Investigator — University at Buffalo; Thomas Mariani, PhD, Principal Investigator — University of Rochester
Locations (2):
- United States (2):
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York

REFERENCES:
- [Background] Maitre NL, Ballard RA, Ellenberg JH, Davis SD, Greenberg JM, Hamvas A, Pryhuber GS; Prematurity and Respiratory Outcomes Program. Respiratory consequences of prematurity: evolution of a diagnosis and development of a comprehensive approach. J Perinatol. 2015 May;35(5):313-321. doi: 10.1038/jp.2015.19. Epub 2015 Mar 26. PMID 25811285
- [Background] Pryhuber GS, Maitre NL, Ballard RA, Cifelli D, Davis SD, Ellenberg JH, Greenberg JM, Kemp J, Mariani TJ, Panitch H, Ren C, Shaw P, Taussig LM, Hamvas A; Prematurity and Respiratory Outcomes Program Investigators. Prematurity and respiratory outcomes program (PROP): study protocol of a prospective multicenter study of respiratory outcomes of preterm infants in the United States. BMC Pediatr. 2015 Apr 10;15:37. doi: 10.1186/s12887-015-0346-3. PMID 25886363
- [Background] Scheible KM, Emo J, Yang H, Holden-Wiltse J, Straw A, Huyck H, Misra S, Topham DJ, Ryan RM, Reynolds AM, Mariani TJ, Pryhuber GS. Developmentally determined reduction in CD31 during gestation is associated with CD8+ T cell effector differentiation in preterm infants. Clin Immunol. 2015 Dec;161(2):65-74. doi: 10.1016/j.clim.2015.07.003. Epub 2015 Jul 29. PMID 26232733
- [Result] Misra R, Shah S, Fowell D, Wang H, Scheible K, Misra S, Huyck H, Wyman C, Ryan RM, Reynolds AM, Mariani T, Katzman PJ, Pryhuber GS. Preterm cord blood CD4(+) T cells exhibit increased IL-6 production in chorioamnionitis and decreased CD4(+) T cells in bronchopulmonary dysplasia. Hum Immunol. 2015 May;76(5):329-338. doi: 10.1016/j.humimm.2015.03.007. Epub 2015 Mar 20. PMID 25797206
- [Result] Grier A, Qiu X, Bandyopadhyay S, Holden-Wiltse J, Kessler HA, Gill AL, Hamilton B, Huyck H, Misra S, Mariani TJ, Ryan RM, Scholer L, Scheible KM, Lee YH, Caserta MT, Pryhuber GS, Gill SR. Impact of prematurity and nutrition on the developing gut microbiome and preterm infant growth. Microbiome. 2017 Dec 11;5(1):158. doi: 10.1186/s40168-017-0377-0. PMID 29228972
- [Derived] Hoover J, Wambach J, Vachharajani A, Warner B, Carroll JL, Kemp JS. Postmenstrual age at discharge in premature infants with and without ventilatory pattern instability. J Perinatol. 2020 Jan;40(1):157-162. doi: 10.1038/s41372-019-0530-7. Epub 2019 Oct 14. PMID 31611617